CLINICAL TRIAL: NCT04259944
Title: Post-surgical Liquid Biopsy-guided Treatment of Stage III and High-risk Stage II Colon Cancer Patients: the PEGASUS Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IFOM ETS - The AIRC Institute of Molecular Oncology (Other)
Collaborators: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFOM-CPT005/2019/PO004; 2019-002074-32 (EudraCT Number)
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Colon Cancer
Keywords: liquid biopsy; colon cancer; adjuvant treatment; ctDNA; colorectal cancer; CAPOX; FOLFIRI; CAPE
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Capecitabine; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liquid Biopsy-Guided Adjuvant Treatment (Experimental): A post-surgical LB executed 2-4 weeks after surgery will guide a "Molecular Adjuvant" treatment:
  * ctDNA+ patients: CAPOX for 3 months
  * ctDNA- patients: capecitabine (CAPE) for 6 months. LB after 1 cycle and if found ctDNA+ will be switched to CAPOX.
  A post-Molecular Adjuvant treatment LB will be performed and instruct subsequent treatment:
  * ctDNA+/+ patients: up-scale to a "Molecular Metastatic" treatment with FOLFIRI for 6 months or until radiological progression or toxicity;
  * ctDNA-/+ patients: up-scale to a "Molecular Metastatic" treatment with CAPOX for 6 months or until radiological progression or toxicity. LB after 3 months at the end of treatment and in case of positivity switch to FOLFIRI.
  * ctDNA+/- patients: de-escalate treatment to CAPE for 3 months. 3 LB performed within 3 months and in case of positivity switch to FOLFIRI.
  * ctDNA-/- patients: interventional follow-up comprising 2 further LB and in case of positivity switch to CAPOX treatment.
  Interventions: Drug: CAPOX; Drug: Capecitabine; Drug: FOLFIRI

INTERVENTIONS:
Drug: CAPOX — DAY 1
  * OXA 130 mg/m2 administered as intravenous infusion over 2 hours in 250 mL dextrose 5%
  * CAPE 1000 mg/m2 administrated per os twice daily
  DAY 2-14
  • CAPE 1000 mg/m2 os twice daily
  Cycle length is 3 weeks comprising 2 hours of oxaliplatin infusion every 21 days, 14 days of oral capecitabine and 7 days of resting.
Drug: Capecitabine — DAY 1-14
  • CAPE 1250 mg/m2 os twice daily
  Cycle length is 3 weeks comprising 14 days of oral capecitabine and 7 days of resting.
Drug: FOLFIRI — Day 1:
  * IRI, 180 mg/m2 administered as iv infusion over 30-90 minutes in 250 mL dextrose 5%, concurrently (via a Y-connector) with
  * LV, 400 mg/m2 administered as an iv infusion over 2 hours, in 250 mL dextrose 5%, followed by
  * 5-FU, 400 mg/m2 administered as a bolus injection (iv push administered by hand) and then at 2400 mg/m2 administered as a iv infusion over 46 hours.
  Cycle length is 2 weeks comprising approximately 48 hours of infusion and 12 days of rest.

SUMMARY:
PEGASUS is a prospective multi-centric study designed to prove the feasibility of using liquid biopsy to guide the post-surgical and post-adjuvant clinical management in 140 microsatellite stable Stage-III and T4N0 Stage-II colon cancer patients.

DETAILED DESCRIPTION:
The LUNAR1 Test (Guardant Health, Redwood City, CA, USA) will be used for ctDNA determination. For the efficacy analysis, the PEGASUS cohort will be compared with a cohort of 420 patients from the TOSCA trial (NCT00646607) population matched 3:1 for all known prognostic phenotypes.

A post-surgical LB executed 2-4 weeks after surgery will guide a "Molecular Adjuvant" treatment as follows: i) ctDNA+ patients will receive CAPOX for 3 months; ii) ctDNA- patients will receive capecitabine (CAPE) for 6 months but will be retested after 1 cycle, and if found ctDNA+ will be switched to CAPOX treatment.

Immediately after the end of the "Molecular Adjuvant" treatment a further LB will be performed and instruct subsequent treatment. Positive patients (ctDNA+/+ and ctDNA-/+) will receive an up-scaled "Molecular Metastatic" systemic treatment for 6 months or until radiological progression or toxicity as follows: i) ctDNA+/+ patients will be treated with FOLFIRI; ii) ctDNA-/+ patients with CAPOX. These patients will be subjected to a LB after 3 months at the end of treatment and in case of positivity will be switched to FOLFIRI.

Patients experiencing ctDNA conversion to negative (ctDNA+/-) will receive a de-escalated treatment with CAPE for 3 months. 3 LB will be performed within 3 months and in case of positivity the patient will be switched to FOLFIRI. Patients with ctDNA-/- will be subjected to an interventional follow-up comprising 2 further LB and in case of positivity they will be switched to CAPOX treatment. PEGASUS is piggybacked to AlfaOmega (NCT04120935), a Master Observational Protocol that will follow patients from diagnosis to 5 years or recurrence/death (whichever comes first), collecting clinical data, radio-images and biological samples. AlfaOmega provides a clinical and logistic ecosystem for the seamless integration of PEGASUS clinical results with the biological underpinning of colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pegasus trial written informed consent.
* Age ≥ 18 years.
* Histologically confirmed diagnosis of operable stage III or T4N0 stage II colon cancer located 12 cm from the anal verge by endoscopy and above the peritoneal reflection at surgery.
* Availability of plasma collected prior to surgery.
* Availability of the original FFPE tumor tissue.
* Acceptance to undergo at least all the interventional liquid biopsies.
* ECOG performance status 0-1.
* Normal organ functions. (as defined in section 9.3)
* Women with childbearing potential should complete a pregnancy test and be willing to use highly effective contraceptive methods.

Exclusion Criteria:- Patients having a MSI-H/MMRd tumor are excluded from the study (done according to standard clinical practice).

* History of another neoplastic disease, unless in remission for ≥ 5 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Had an incomplete diagnostic colonoscopy and/or polyps removal.
* Macroscopic or microscopic evidence of residual tumor (R1 or R2 resections). Patients should never have had any evidence of metastatic disease (including presence of tumor cells in the peritoneal lavage).
* Current or recent treatment with another investigational drug or participation in another investigational study
* Patient unable to comply with the study protocol owing to psychological, social or geographical reasons.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Inadequate contraception (male or female patients) if of childbearing or procreational potential.
* Clinically relevant cardiovascular disease.
* Acute or subacute intestinal occlusion or history of inflammatory bowel disease.
* Pre-existing neuropathy > grade 1. Known grade 3 or 4 allergic reaction to any of the components of the treatment.
* Has a known DPD (DihydroPyrimidine Dehydrogenase) deficiency.
* Has a known Gilbert Syndrome or UGT1A1 homozygous *28/*28 germline variant.
* Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Number of post-surgery and post-adjuvant false negative cases after a double ctDNA-negative detection | 2 years
  Cases that become positive at subsequent interventional LB or that experience radiological relapse

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | 2 & 3 years
Overall Survival (OS) | 5 years
Safety and tolerability according to CTCAE version 5.0 | 2 years
Assessment of QLQ-C30 and CR-29 EORTC questionnaires | 2 years
Number of patients experiencing ctDNA seroconversion (i.e. ctDNA+ that become ctDNA-) after any chemotherapy regimen remaining disease free | 2 & 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lonardi, MD, Study Chair — Istituto Oncologico Veneto IRCCS
Locations (11):
- Italy (7):
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Niguarda Cancer Center, ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
  - Ospedale Santa Maria della Misericordia, Perugia
  - AULS della Romagna, Ravenna
- Spain (4):
  - Hospital Moises Broggi, Sant Joan Despí, Barcelona
  - University Hospital del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology, Barcelona
  - INCLIVA Biomedical Research Institute, Valencia